CLINICAL TRIAL: NCT04799340
Title: Characterizing and Remediating Recollection-specific Face Recognition Deficits in Developmental Prosopagnosia
Brief Title: Computer-based Training of Face Recollection to Improve Face Recognition in Developmental Prosopagnosia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston VA Research Institute, Inc. (Other)
Responsible Party: Principal Investigator, Joseph DeGutis, Assistant Professor, Harvard Medical School (HMS and HSDM)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21EY031000, R01EY032510; R21EY031000 (NIH)
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Developmental Prosopagnosia
MeSH Terms: conditions — Prosopagnosia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- holistic face training + repetition lag training (Experimental)
  Interventions: Behavioral: cognitive training
- waitlist control (No Intervention)

INTERVENTIONS:
Behavioral: cognitive training — training to improve encoding and recognition of faces
  Arms: holistic face training + repetition lag training

SUMMARY:
This study will examine the effectiveness of a cognitive training intervention targeting face recollection, repetition lag training, at improving face recognition in Developmental Prosopagnosia.

ELIGIBILITY:
Inclusion Criteria:

Developmental prosopagnosic participants will be included if they are...

* aged 18-90,
* have lifelong histories of face recognition difficulties that impact their everyday life (i.e., not associated with some event such as a stroke, seizure, etc)
* score significantly below the mean on the famous faces test and Cambridge Face Memory Test

Exclusion Criteria:

Participants will be excluded from the study if they...

* have a history of a significant neurological disorder including hydrocephalus, stroke, moderate to severe traumatic brain injury (TBI), severe neuromuscular diseases, or severe hypoxia due to cardiac arrest.
* have impairments that interfere with cognitive performance, such as uncorrected hearing or vision, lack of English proficiency, musculoskeletal or other issues
* have psychiatric disorders, such as schizophrenia, major depressive disorder, bipolar disorder, chronic intractable obsessive-compulsive disorder, or agoraphobia.
* We will exclude individuals who are currently dependent on alcohol or other substances, as this may negatively impact cognitive performance.
* We will exclude participants who currently are, or within the last 6 months, participating in a behavioral or pharmacological intervention.
* Patients with a history of mild TBI or simple concussion will not be excluded as long as it was > 6 months ago and as long as they have not had repeated concussions (>5)
* We will include individuals with a diagnosis of ADHD as long as their medication has been consistent for the past 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Cambridge Face Memory Test | 15 minutes
  learning and recognizing novel faces, out of 72 (higher score is better)
Face Recollection | 15 minutes
  old/new face recognition test, extracting familiarity and recollection parameters, higher score is better
Face Perception | 30 minutes
  composite of face matching tasks, Cambridge Face perception Test and computerized Benton, higher score is better

SECONDARY OUTCOMES:
Self-reported face recognition | 5 minutes
  questionnaire
Face-name learning task | 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- VA Boston Healthcare System, 150 S. Huntington Ave., Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided